CLINICAL TRIAL: NCT00484198
Title: A Randomized, Double-blind, Placebo and Active Comparator-Controlled, Parallel-Group Study of the Efficacy and Safety of Rivoglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Brief Title: Study of Rivoglitazone in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS0011-A-U301; 2006-005047-28 (EudraCT Number)
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; rivoglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental): Rivoglitazone 1.0 mg
  Interventions: Drug: Rivoglitazone
- 3 (Experimental): Rivoglitazone 1.5 mg
  Interventions: Drug: Rivoglitazone
- 4 (Active Comparator): Pioglitazone 45 mg
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — 45 mg over-encapsulated tablet administered orally, once daily
  Other Names: Actos
  Arms: 4
Drug: Placebo — Rivoglitazone-matching placebo administered as a tablet orally, once daily or a pioglitazone-matching placebo administered as an over-encapsulated tablet orally, once daily capsule
  Arms: 1
Drug: Rivoglitazone — 1.0 mg tablet administered orally, once daily
  Arms: 2
Drug: Rivoglitazone — 1.5 mg tablet administered orally, once daily
  Arms: 3

SUMMARY:
This is a 26-week study in subjects with type 2 diabetes currently sub-optimally controlled by diet and exercise or with non-thiazolidinedione antihyperglycemic monotherapy. The total duration of a subject's participation will be approximately 30 weeks, including a 2-week placebo run-in period, a 26-week double-blind treatment period, and a 2-week post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Male or female at least 18 years of age
* Hemoglobin A1C > 7% and less or equal to 8.5%
* Non-fasting C-peptide > 0.5 ng/mL
* Current monotherapy treatment with stable dose of approved non-Thiazolidinedione (TZD) antihyperglycemic medication for greater or equal to 3 months prior to screening or
* Untreated with any antihyperglycemic agent during 2 months prior to screening

Exclusion Criteria:

* History of type 1 diabetes or ketoacidosis
* History of long-term therapy with insulin
* Body Mass Index (BMI) > 45 kg/m^2
* Known history of Congestive Heart Failure (CHF)
* Impaired hepatic function
* History of prior treatment failure with, or intolerance of, a TZD
* Contraindication to treatment with pioglitazone
* Treatment with fibrates
* If untreated with oral antihyperglycemic, considered to have failed diet and exercise modification as the sole treatment for type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1912 (Actual)
Dates: Start 2007-04-23 (Actual); Primary Completion 2009-02-12 (Actual); Study Completion 2009-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (183):
- United States (70):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Hoover, Alabama
  - Muscle Shoals, Alabama
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Buena Park, California
  - Garden Grove, California
  - Huntington Park, California
  - Los Angeles, California
  - Paramount, California
  - Sacramento, California
  - San Diego, California
  - Walnut Creek, California
  - West Covina, California
  - West Hills, California
  - Denver, Colorado
  - Delray Beach, Florida
  - Jacksonville, Florida
  - Merritt Island, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Honolulu, Hawaii
  - Boise, Idaho
  - Chicago, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Madisonville, Kentucky
  - New Orleans, Louisiana
  - Slidell, Louisiana
  - Springfield, Massachusetts
  - Portage, Michigan
  - Southfield, Michigan
  - St Louis, Missouri
  - Voorhees Township, New Jersey
  - Syracuse, New York
  - Morehead City, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Delaware, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Cleveland, Tennessee
  - Kingsport, Tennessee
  - New Tazewell, Tennessee
  - Carrollton, Texas
  - Conroe, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Garland, Texas
  - Irving, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Olympia, Washington
  - Milwaukee, Wisconsin
- Argentina (3):
  - Loma Verde, Buenos Aires
  - Zárate, Buenos Aires
  - San Vicente, Córdoba Province
- Austria (3):
  - Feldkirch
  - Graz
  - Vienna
- Chile (3):
  - Santiago, Providencia
  - Santiago
  - Temuco
- Czechia (7):
  - Horní Město
  - Karlovy Vary
  - Prague
  - Ústí nad Labem
  - Vysoký Les
  - Zlín
  - Znojmo
- Germany (19):
  - Aschaffenburg
  - Augsburg
  - Bad Oeynhausen
  - Berlin
  - Bosenheim
  - Dortmund
  - Dresden
  - Friedrichsthal
  - Giessen
  - Halle
  - Hamburg
  - Kippenheim
  - Mainz
  - Rehlingen
  - Riesa
  - Saarbrücken
  - Saarlouis
  - Siegen
  - Wiesbaden
- Hungary (8):
  - Balatonfüred
  - Békéscsaba
  - Budapest
  - Debrecen
  - Eger
  - Gyula
  - Kaposvár
  - Szentes
- India (21):
  - Hyderabad, Andhra Pradesh
  - Vijayawada, Andhra Pradesh
  - Visakhapatnam, Andhra Pradesh
  - Vasanth Nagar, Bangalore
  - Mylapore, Chennai
  - Shāstri Nagar, Ghaziabad
  - Ahmedabad, Gujarat
  - Gandhinagar, Gujarat
  - Karnāl, Haryana
  - Sarwa C., Jaipur
  - Bangalore, Karnataka
  - Belagavi, Karnataka
  - Mangalore, Karnataka
  - Kochi, Kerala
  - Indore, Madhya Pradesh
  - Mumbai, Maharashtra
  - Dhantoli, Nagpur
  - Rāmdaspeth, Nagpur
  - Jaipur, Rajasthan
  - Coimbatore, Tamil Nadu
  - Aligarh, Uttar Pradesh
- Latvia (4):
  - Daugavpils
  - Kuldīga
  - Liepāja
  - Riga
- Mexico (7):
  - Cuernavaca, Morelos
  - Monterrey, Nuevo León
  - Metepec, Toluca
  - Mérida, Yucatán
  - Aguascalientes
  - Durango
  - Puebla City
- Peru (6):
  - La Victoria, Lima region
  - Magdalena del Mar, Lima region
  - San Juan de Miraflores, Lima region
  - San Martín de Porres, Lima region
  - Monterrico, Sucro Lima
  - Lima
- Puerto Rico (3):
  - Villa Fontana, Carolina
  - Rio Piedras
  - San Juan
- Romania (5):
  - Arad
  - Brasov
  - Bucharest
  - Satu Mare
  - Târgu Mureş
- Serbia (5):
  - Belgrade
  - Kragujevac
  - Niš
  - Subotica
  - Zemun
- Slovakia (6):
  - Bratislava
  - Lučenec
  - Moldava nad Bodvou
  - Nové Mesto nad Váhom
  - Považská Bystrica
  - Žilina
- South Africa (2):
  - Johannesburg
  - Port Elizabeth
- Ukraine (5):
  - Dnipro
  - Kharkiv
  - Kiev
  - Lviv
  - Simferopol
- United Kingdom (6):
  - Edmonton, London
  - Sunbury-on-Thames, Middlesex
  - Addlestone, Surrey
  - Wakefield, West Yorks
  - Swindon, Wiltshire
  - Chippenham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1,912 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 254 sites in Africa, Asia, Europe, North America, and South America.
Pre-assignment Details: During the 2-week stabilization/washout, single-blind, placebo run-in period, participants were to discontinue any previous therapy with oral anti-hyperglycemic agents and were to self-administer single-blind, double-dummy, placebo medication consisting of over-encapsulated pioglitazone-matching placebo tablets and rivoglitazone-matching placebo tablets once daily.
Groups:
- Placebo: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone-matching placebo tablet or a Pioglitazone-matching placebo over-encapsulated tablet once daily for 26 weeks.
  Extension Period:
  Participants who received Placebo in the base study received Pioglitazone 45 mg once daily for 26-week cycles (Cycle 1 and 2) instead in the extension period.
- Rivoglitazone 1.0 mg: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone 1.0 mg tablet once daily for 26 weeks.
  Extension Period:
  Participants with type 2 diabetes mellitus who were administered a Rivoglitazone 1.0 mg tablet once daily for 26 week cycles (Cycle 1 and 2).
- Rivoglitazone 1.5 mg: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone 1.5 mg tablet once daily for 26 weeks.
  Extension Period:
  Participants with type 2 diabetes mellitus who were administered a Rivoglitazone 1.5 mg tablet once daily for 26 weeks cycles (Cycle 1 and 2).
- Pioglitazone 45 mg: Participants with type 2 diabetes mellitus who were administered a Pioglitazone 45 mg over-encapsulated tablet once daily for 26 weeks.
  Extension Period:
  Participants with type 2 diabetes mellitus who were administered a Pioglitazone 45 mg over-encapsulated tablet once daily for 26 week cycles (Cycle 1 and Cycle 2).
Period: Overall Study
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5 mg | Pioglitazone 45 mg
Started | 137 | 274 | 750 | 751
Completed | 96 | 208 | 599 | 579
Not Completed | 41 | 66 | 151 | 172
Not completed — Participant Withdrew Consent | 12 | 21 | 47 | 59
Not completed — Hyperglycemia Meeting Discontinuation Criteria | 16 | 17 | 29 | 38
Not completed — Therapeutic failure/ lack of efficacy | 3 | 2 | 6 | 8
Not completed — Adverse Event | 3 | 11 | 32 | 31
Not completed — Protocol Violation | 0 | 5 | 6 | 8
Not completed — Other | 7 | 10 | 31 | 28

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the All Randomized set.
Groups:
- Placebo: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone-matching placebo tablet or a Pioglitazone-matching placebo over-encapsulated tablet once daily for 26 weeks.
- Rivoglitazone 1.0 mg: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone 1.0 mg tablet once daily for 26 weeks.
- Rivoglitazone 1.5 mg: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone 1.5 mg tablet once daily for 26 weeks.
- Pioglitazone 45 mg: Participants with type 2 diabetes mellitus who were administered a Pioglitazone 45 mg over-encapsulated tablet once daily for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5 mg | Pioglitazone 45 mg | Total
Number analyzed (Participants) | 137 | 274 | 750 | 751 | 1912
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.32) | 55.0 (10.51) | 55.1 (10.59) | 55.0 (10.84) | 55.0 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 142 | 368 | 353 | 933
  Male | 67 | 132 | 382 | 398 | 979
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 59 | 171 | 151 | 414
  Not Hispanic or Latino | 104 | 215 | 579 | 600 | 1498
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 11 | 1 | 17
  Asian | 42 | 89 | 245 | 243 | 619
  Black or African American | 2 | 17 | 33 | 35 | 87
  White | 80 | 147 | 406 | 414 | 1047
  Other | 11 | 18 | 55 | 58 | 142

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c at Baseline and Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Percentage of hemoglobin A1c (HbA1c) levels are reported.
Time Frame: Baseline up to week 26 post-dose
Population: Hemoglobin A1c (HbA1c) levels were assessed using the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Groups:
- Rivoglitazone 1.5mg: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone 1.5 mg tablet once daily for 26 weeks.
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 134 | 266 | 733 | 728
percentage of HbA1c
  Baseline | 7.7 (0.55) | 7.7 (0.54) | 7.7 (0.57) | 7.7 (0.58)
  Week 26 | 8.0 (0.86) | 7.3 (0.94) | 7.1 (0.83) | 7.2 (0.90)

2. Primary Outcome: Change in Hemoglobin A1c From Baseline Through Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Percent change in hemoglobin (HbA1c) levels are reported. Greater (negative) percent change indicates improvement.
Time Frame: Baseline up to 26 weeks post-dose
Population: Change in hemoglobin A1c (HbA1c) levels were assessed using the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percent change in HbA1c
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 134 | 266 | 733 | 728
percent change in HbA1c | 0.3 (0.69) | -0.3 (0.75) | -0.6 (0.72) | -0.5 (0.77)

3. Secondary Outcome: Fasting Plasma Glucose From Baseline Through Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Normal fasting plasma glucose (FPG) levels are being reported. Normal FPG levels range from 70-110 mg/dL. Lower FPG values indicates better clinical outcome, ie. improvement in FPG.
Time Frame: Baseline up to week 26 post-dose
Population: Fasting plasma glucose levels were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 133 | 263 | 729 | 721
mg/dL
  Baseline | 161.1 (44.28) | 159.2 (42.33) | 160.9 (40.24) | 161.9 (42.96)
  Week 26 | 167.5 (41.23) | 136.5 (39.73) | 128.6 (35.06) | 132.3 (38.32)

4. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline Through Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: The change in normal fasting plasma glucose (FPG) levels are being reported. A greater (negative) change from baseline indicates an improvement in FPG.
Time Frame: Baseline up to 26 weeks post-dose
Population: Change in fasting plasma glucose levels were assessed in participants with values at both baseline and study endpoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 133 | 263 | 729 | 721
mg/dL | 6.1 (39.61) | -22.1 (34.75) | -32.4 (38.48) | -29.5 (40.32)

5. Secondary Outcome: Homeostasis Model Assessment Index for Insulin Resistance At Baseline To Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Homeostasis Model Assessment index for Insulin Resistance (HOMA-IR) was calculated as:
  (fasting insulin concentration [μU/mL] x fasting glucose concentration [mmol/L])/22.5 Low HOMA-IR scores indicate high insulin sensitivity, whereas high HOMA-IR scores indicate low insulin sensitivity (insulin resistance). A normal HOMA-IR score is <2.60, HOMA-IR scores 2.60-3.80 are considered "borderline high", and HOMA-IR scores >3.80 are considered "high" and have correlations of insulin resistance. High HOMA-IR scores indicate worse outcome.
Time Frame: Baseline up to week 26 post-dose
Population: Homeostasis Model Assessment Index was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 104 | 243 | 690 | 671
score on a scale
  Baseline | 6.2 (6.98) | 5.6 (4.64) | 6.0 (6.65) | 6.2 (6.92)
  Week 26 | 6.8 (5.65) | 4.0 (3.78) | 3.7 (4.49) | 4.1 (4.75)

6. Secondary Outcome: Change in Homeostasis Model Assessment Index for Insulin Resistance At Baseline To Week 26 Endpoint With Last Observation Carried Forward Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: The change in the Homeostasis Model Assessment index for Insulin Resistance (HOMA-IR) was calculated as:
  (fasting insulin concentration [μU/mL] x fasting glucose concentration [mmol/L])/22.5 Low HOMA-IR scores indicate high insulin sensitivity, whereas high HOMA-IR scores indicate low insulin sensitivity (insulin resistance). A normal HOMA-IR score is <2.60, HOMA-IR scores 2.60-3.80 are considered "borderline high", and HOMA-IR scores >3.80 are considered "high" and have correlations of insulin resistance. A negative HOMA-IR score indicates an improvement in insulin sensitivity.
Time Frame: Baseline up to 26 weeks post-dose
Population: Change in Homeostasis Model Assessment Index was assessed in participants with values for baseline and study endpoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 104 | 243 | 690 | 671
score on a scale | 0.4 (7.56) | -1.5 (3.79) | -2.3 (5.15) | -2.2 (7.56)

7. Secondary Outcome: Total Cholesterol At Baseline To Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Total cholesterol is a measure of the total amount of cholesterol in the blood, including low-density lipoprotein cholesterol (LDL-C) - the "bad" cholesterol, high-density lipoprotein cholesterol (HDL-C) - the "good" cholesterol, and triglycerides. The equation to calculate total cholesterol is: LDL + HDL + (triglycerides/5) = total cholesterol.
Time Frame: Baseline up to week 26 post-dose
Population: Total cholesterol levels were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 106 | 246 | 694 | 678
mg/dL
  Baseline | 190.1 (36.23) | 193.4 (38.27) | 191.6 (38.80) | 189.8 (39.42)
  Week 26 | 191.9 (39.60) | 198.0 (40.39) | 199.1 (43.14) | 194.6 (41.84)

8. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Total cholesterol is a measure of the total amount of cholesterol in the blood, including low-density lipoprotein cholesterol (LDL-C) - the "bad" cholesterol, high-density lipoprotein cholesterol (HDL-C) - the "good" cholesterol, and triglycerides. The equation to calculate total cholesterol is: LDL + HDL + (triglycerides/5) = total cholesterol. Higher percent change in total cholesterol indicates better outcome, ie. improvement.
Time Frame: Baseline up to 26 weeks post-dose
Population: Percent change in total cholesterol levels were assessed in participants with values at baseline and study endpoint.
Measure: Mean (Standard Deviation); unit: percent change in total cholesterol
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 106 | 246 | 694 | 678
percent change in total cholesterol | 1.9 (13.01) | 4.0 (17.81) | 5.3 (17.49) | 3.6 (16.31)

9. Secondary Outcome: Total Triglycerides At Baseline To Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Total Triglycerides (TG) is a measure of the total amount of triglycerides in the blood. The equation to calculate total triglycerides is: (total cholesterol-Low-density Lipoprotein cholesterol (LDL- C) - High-density lipoprotein cholesterol (HDL- C)) x 5 = Total Triglycerides. Normal triglyceride levels are below 150 mg/dL.
Time Frame: Baseline up to Week 26 post-dose
Population: Total triglyceride levels were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 106 | 246 | 694 | 678
mg/dL
  Baseline | 185.6 (111.25) | 173.3 (104.90) | 169.5 (101.27) | 175.0 (96.75)
  Week 26 | 170.5 (99.17) | 148.0 (91.88) | 141.0 (84.12) | 152.1 (112.72)

10. Secondary Outcome: Percent Change in Total Triglycerides From Baseline to Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Total Triglycerides (TG) is a measure of the total amount of triglycerides in the blood. The equation to calculate total triglycerides is: (total cholesterol-Low-density Lipoprotein cholesterol (LDL- C) - High-density lipoprotein cholesterol (HDL- C)) x 5 = Total Triglycerides. A negative change means better outcome, ie. improvement.
Time Frame: Baseline up to 26 weeks post-dose
Population: Percent change in total triglyceride levels were assessed in participants with values at baseline and study endpoint.
Measure: Mean (Standard Deviation); unit: percent change in total triglycerides
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 106 | 246 | 694 | 678
percent change in total triglycerides | -1.8 (26.52) | -10.3 (32.84) | -11.7 (34.35) | -9.6 (45.84)

11. Secondary Outcome: Low-Density Lipoprotein Cholesterol At Baseline To Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Low-density lipoprotein cholesterol (LDL-C), "bad" cholesterol, is a measure of the total amount of low-density lipoprotein cholesterol in the blood. Normal LDL levels are <100 mg/dL.
Time Frame: Baseline up to Week 26 post-dose
Population: Low-density lipoprotein cholesterol levels were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 106 | 246 | 694 | 674
mg/dL
  Baseline | 108.5 (29.68) | 112.8 (32.37) | 112.1 (32.35) | 110.5 (33.60)
  Week 26 | 111.8 (31.37) | 118.0 (34.19) | 118.7 (36.99) | 115.0 (36.03)

12. Secondary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol From Baseline to Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Low-density lipoprotein cholesterol (LDL-C), "bad" cholesterol, is a measure of the total amount of low-density lipoprotein cholesterol in the blood. A higher percent change indicates improvement.
Time Frame: Baseline up to 26 weeks post-dose
Population: Percent change in low-density lipoprotein cholesterol was assessed in participants with values at baseline and study endpoint.
Measure: Mean (Standard Deviation); unit: percent change in LDL
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 106 | 246 | 694 | 674
percent change in LDL | 3.4 (18.56) | 9.3 (32.91) | 9.6 (30.02) | 7.3 (32.25)

13. Secondary Outcome: High-Density Lipoprotein Cholesterol At Baseline To Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: High-density lipoprotein cholesterol (HDL-C), "good" cholesterol, is a measure of the total amount of high-density lipoprotein cholesterol in the blood. Normal HDL levels are >40 mg/dL.
Time Frame: Baseline to Week 26 post-dose
Population: High-density lipoprotein cholesterol was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 106 | 246 | 694 | 675
mg/dL
  Baseline | 45.3 (11.73) | 46.0 (12.49) | 45.8 (11.46) | 44.7 (10.25)
  Week 26 | 45.6 (11.46) | 50.4 (14.84) | 52.0 (14.72) | 49.7 (12.65)

14. Secondary Outcome: Percent Change in High-Density Lipoprotein Cholesterol From Baseline to Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: High-density lipoprotein cholesterol (HDL-C), "good" cholesterol, is a measure of the total amount of high-density lipoprotein cholesterol in the blood. A higher percent change indicates improvement.
Time Frame: Baseline to 26 weeks post-dose
Population: Percent change in high-density lipoprotein cholesterol was assessed in participants with values at baseline and study endpoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 106 | 246 | 694 | 675
percent change | 2.7 (14.30) | 10.3 (18.15) | 14.8 (22.65) | 12.3 (21.97)

15. Secondary Outcome: Apolipoprotein A-I At Baseline To Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Apolipoprotein (Apo) A-I levels, a measure of the total amount of Apolipoprotein (Apo) A-I in the blood, are being reported. Normal Apo A-1 levels range from 120-140 mg/dL.
Time Frame: Baseline to Week 26 post-dose
Population: Apolipoprotein A-I was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 105 | 245 | 691 | 677
mg/dL
  Baseline | 145.3 (25.11) | 145.7 (27.60) | 145.2 (24.31) | 143.6 (22.88)
  Week 26 | 146.2 (26.39) | 146.4 (29.52) | 145.9 (27.37) | 143.9 (24.97)

16. Secondary Outcome: Percent Change in Apolipoprotein A-I From Baseline to Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Apolipoprotein (Apo) A-I is a measure of the total amount of Apolipoprotein (Apo) A-I in the blood. Decreased ApoA-1 levels are associated with poor clinical outcome. A lower percent change in ApoA-1 levels indicates an improvement in clinical outcome.
Time Frame: Baseline up to 26 weeks post-dose
Population: Percent change in apolipoprotein A-I was assessed in participants with values at baseline and study endpoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 105 | 245 | 691 | 677
percent change | 2.0 (12.22) | 1.0 (12.88) | 0.9 (13.18) | 0.8 (13.09)

17. Secondary Outcome: Apolipoprotein B At Baseline To Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Apolipoprotein (Apo) B, a measure of the total amount of Apo B in the blood, is being reported. Normal Apo B levels are <100 mg/dL.
Time Frame: Baseline to Week 26 post-dose
Population: Apolipoprotein B was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 105 | 245 | 691 | 677
mg/dL
  Baseline | 112.8 (25.24) | 116.1 (26.49) | 114.6 (26.88) | 114.3 (27.33)
  Week 26 | 115.3 (26.50) | 113.6 (28.60) | 111.5 (30.29) | 110.3 (28.90)

18. Secondary Outcome: Percent Change in Apolipoprotein B From Baseline to Week 26 Endpoint With Last Observation Carried Forward (LOCF) Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Apolipoprotein (Apo) B, a measure of the total amount of Apo B in the blood, is being reported. A greater (negative) percent change in ApoB levels indicated an improvement in clinical outcome.
Time Frame: Baseline up to 26 weeks post-dose
Population: Apolipoprotein B was assessed in participants with values at baseline and study endpoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 105 | 245 | 691 | 677
percent change | 3.0 (14.83) | -0.4 (19.46) | -1.1 (21.24) | -2.5 (18.17)

19. Secondary Outcome: Hemoglobin A1c at Baseline and Week 52 Extension Period Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Percentage of hemoglobin A1c (HbA1c) levels are reported.
Time Frame: Baseline up to Week 52 post-dose
Population: Hemoglobin A1c levels were assessed using the Study Extension Set.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Groups:
- Placebo/Pioglitazone 45 mg: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone-matching placebo tablet or a Pioglitazone-matching placebo over-encapsulated tablet once daily for 26 weeks.
Arm/Group | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg | Placebo/Pioglitazone 45 mg
Number analyzed (Participants) | 66 | 200 | 194 | 27
percentage of HbA1c
  Baseline | 7.5 (0.46) | 7.6 (0.53) | 7.6 (0.51) | 7.4 (0.48)
  Week 52: number analyzed (Participants) | 27 | 65 | 54 | 11
  Week 52 | 7.0 (0.72) | 6.9 (0.60) | 6.9 (0.58) | 7.0 (0.75)

20. Secondary Outcome: Change in Hemoglobin A1c From Baseline Through Week 52 Extension Period Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Change in hemoglobin (HbA1c) levels are reported. Greater (negative) percent change indicates improvement.
Time Frame: Baseline up to 52 weeks post-dose
Population: Hemoglobin A1c was assessed in participants with values at baseline and the extension visit at the end of Cycle 1.
Measure: Mean (Standard Deviation); unit: percent change in HbA1c
Groups:
- Placebo/ Pioglitazone 45 mg: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone-matching placebo tablet or a Pioglitazone-matching placebo over-encapsulated tablet once daily for 26 weeks.
Arm/Group | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg | Placebo/ Pioglitazone 45 mg
Number analyzed (Participants) | 27 | 65 | 54 | 11
percent change in HbA1c | -0.5 (0.69) | -0.7 (0.57) | -0.7 (0.67) | -0.4 (0.70)

21. Secondary Outcome: Fasting Plasma Glucose From Baseline Through Week 52 Extension Period Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: as for outcome 3
Time Frame: Baseline up to Week 52 post-dose
Population: Fasting plasma glucose (FPG) levels were assessed in participants with available data in the Study Extension Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg | Placebo/ Pioglitazone 45 mg
Number analyzed (Participants) | 64 | 200 | 193 | 27
mg/dL
  Baseline | 147.4 (32.31) | 152.8 (32.32) | 149.0 (36.00) | 142.5 (27.81)
  Week 52: number analyzed (Participants) | 21 | 48 | 38 | 7
  Week 52 | 117.8 (27.93) | 116.6 (24.12) | 115.6 (19.04) | 124.9 (36.92)

22. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline Through Week 52 Extension Period Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: as for outcome 4
Time Frame: Baseline up to 52 weeks post-dose
Population: Fasting plasma glucose (FPG) was assessed in participants with values at baseline and the extension visit at the end of Cycle 1. Participants who did not have both baseline and Week 52 data were not included in this analysis (n=1 each for Rivoglitazone 1.0 mg and Pioglitazone 45 mg groups).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg | Placebo/ Pioglitazone 45 mg
Number analyzed (Participants) | 20 | 48 | 37 | 7
mg/dL | -33.8 (41.48) | -34.2 (24.86) | -29.5 (31.39) | -35.9 (20.75)

23. Secondary Outcome: Drug-Related Treatment-Emergent Adverse Events Reported by ≥1% Participants Following Rivoglitazone or Pioglitazone Compared to Placebo as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that occurred on or after the first dose of double-blind study medication, and ongoing AEs that started prior to the first dose of double-blind study medication and increased in severity on or after the first dose of double-blind study medication.
Time Frame: Week -2 up to Week 52 post-dose
Population: Drug-related TEAEs were assessed in the Safety Set which included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline safety measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
Number analyzed (Participants) | 137 | 269 | 741 | 739
Participants
  Participants with drug-related TEAEs | 15 | 50 | 144 | 134
  Gastritis | 1 | 3 | 2 | 7
  Edema | 0 | 2 | 5 | 9
  Edema peripheral | 1 | 14 | 46 | 46
  Pitting edema | 0 | 6 | 10 | 13
  Weight increased | 0 | 5 | 23 | 12
  Fluid retention | 0 | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) data were assessed from the signing of the informed consent (Week -2) up to 52 weeks post-dose for the duration of the study period.
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that occurred on or after the first dose of double-blind (DB) study medication, and ongoing AEs that started prior to the first dose of DB study medication and increased in severity on or after the first dose of DB study medication. TEAEs were reported from the Safety Set which included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline safety measurement.
Arm/Group | Placebo | Rivoglitazone 1.0 mg | Rivoglitazone 1.5mg | Pioglitazone 45 mg
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/269 | 0/741 | 2/739
Serious Adverse Events (participants affected / at risk) | 3/137 | 10/269 | 22/741 | 28/739
Other Adverse Events (participants affected / at risk) | 56/137 | 131/269 | 408/741 | 374/739
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=137) | Rivoglitazone 1.0 mg (N=269) | Rivoglitazone 1.5mg (N=741) | Pioglitazone 45 mg (N=739)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 3
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2
Basedow's disease (Endocrine disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hernia obstructive (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Spinal compression (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral ischemia (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Ischemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Status migrainous (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 2 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=137) | Rivoglitazone 1.0 mg (N=269) | Rivoglitazone 1.5mg (N=741) | Pioglitazone 45 mg (N=739)
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 14 | 17
Gastritis (Gastrointestinal disorders) | 3 | 5 | 10 | 9
Edema peripheral (General disorders) | 3 | 18 | 54 | 56
Pitting edema (General disorders) | 0 | 7 | 10 | 17
Bronchitis (Infections and infestations) | 4 | 5 | 24 | 20
Gastroenteritis (Infections and infestations) | 1 | 4 | 15 | 7
Influenza (Gastrointestinal disorders) | 3 | 5 | 15 | 17
Nasopharyngitis (Infections and infestations) | 6 | 13 | 40 | 41
Upper respiratory tract infection (Infections and infestations) | 3 | 8 | 38 | 25
Urinary tract infection (Infections and infestations) | 6 | 19 | 34 | 30
Weight increased (Investigations) | 0 | 5 | 24 | 14
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 1 | 7 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7 | 24 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 19 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4 | 13 | 20
Dizziness (Nervous system disorders) | 1 | 4 | 15 | 7
Headache (Nervous system disorders) | 5 | 7 | 27 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 7 | 10
Hypertension (Vascular disorders) | 4 | 4 | 18 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No